CLINICAL TRIAL: NCT03062878
Title: The Effects of Anthracycline-based Chemotherapy on Spontaneous Baroreflex Sensitivity, Carotid Artery Stiffness, and Endothelial-dependent Vascular Function.
Brief Title: The Effects of Anthracycline-based Chemotherapy on Peripheral Vascular Function
Status: Completed | Type: Observational
Sponsor: Carl Ade, M.S., Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Carl Ade, M.S., Ph.D., Assistant Professor, Kansas State University
Organization: Kansas State University (Other)
Other Study IDs: Pro8425
Record Dates: First submitted 2017-02-16; First posted 2017-02-24 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Lymphoma; Chemotherapy Effect
MeSH Terms: conditions — Breast Neoplasms; Lymphoma | interventions — Arterial Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Breast Cancer/Lymphoma Patient: Breast cancer or lymphoma patients currently undergoing anthracycline-based chemotherapy treatment. Patients are eligible if they have completed at least 1 cycle of chemotherapy. Free of known clinical cardiovascular disease.
  Interventions: Other: Arterial blood pressure; Other: Vascular Ultrasound; Other: Venous blood sample; Other: Skin microcirculatory blood flow
- Breast Cancer/Lymphoma Survivor: Individuals with history of breast cancer or lymphoma (1-5 years removed from last date of chemotherapy) who have a treatment history of anthracycline-based chemotherapy. Free of known clinical cardiovascular disease.
  Interventions: Other: Arterial blood pressure; Other: Vascular Ultrasound; Other: Venous blood sample; Other: Skin microcirculatory blood flow
- Control: Individuals with no history of caner or chemotherapy. Free of known clinical cardiovascular disease
  Interventions: Other: Arterial blood pressure; Other: Vascular Ultrasound; Other: Venous blood sample; Other: Skin microcirculatory blood flow

INTERVENTIONS:
Other: Arterial blood pressure — Continuously monitored for 5-30 minutes via finger photoplesmography
Other: Vascular Ultrasound — Assessment of carotid artery cross sectional area and intima-media thickness. Assessment of brachial artery diameter
Other: Venous blood sample — Evaluation of oxidative stress via serum lipid hydroperoxide
Other: Skin microcirculatory blood flow — Assessed non-invasively in the forearm skin via Laser Doppler flowmetry in response to locally delivered acetylcholine (ACh) and sodium nitroprusside (SNP) via iontophoresis.

SUMMARY:
The overall goal of this project is to determine the effects of anti-cancer chemotherapy on reflex control of blood pressure and vascular function. Recent data have demonstrated that cardiovascular disease-related mortality is the 2nd cause of morbidity and mortality for 7-year cancer survivors treated with chemotherapy. This anti-cancer treatment-mediated cardiotoxicity is a progressive process that begins at the molecular level, progresses to myocardial injury and left ventricular dysfunction, cumulating as heart failure and cardiovascular disease-related mortality. In parallel to these cardiac-specific changes, chemotherapy has also been shown to increase the risk for vascular-related abnormalities. However, the impact of adjuvant treatments on the function and structure of the peripheral vascular system remains poorly understood. With normal aging, two of the most important vascular adaptations to arteries, which strongly contribute to the increased risk of vascular-related and general cardiovascular disease, are an increase in large artery stiffness and dysfunction of the vascular endothelium. Therefore, the overall goal of this project is to determine the effects of anthracycline-based chemotherapy on large and small artery function and structure. The central hypothesis is that this type of cancer therapy results in negative vascular consequences as determined by non-invasive evaluation of spontaneous blood pressure control, carotid artery stiffness, and vascular endothelium-dependent vasodilation.

This observational study is designed to increase our understanding of the vascular changes that occur during and following anti-cancer chemotherapy and provide insight into new methods that will decrease cardiovascular disease risk in those treated for cancer.

DETAILED DESCRIPTION:
Cancer remains one of the leading causes of death in modern society. Breast cancer is a prevalent type of cancer in most societies, but due to increasing rates of detection coupled with advanced therapies, of the ≈230,000 people newly diagnosed each year with breast cancer, approximately 90% are expected to live beyond 5 years. Despite the trend in improved cancer-related morality, cancer survivors are at a significantly increased risk for cardiovascular disease (CVD) morbidity and mortality. As such, approximately $800 million is spent annually in providing cardiovascular care for female cancer survivors alone. In a recent study, Daher et al. (2012) reported a Framingham Risk Score of 8.4 and a 10-year risk of general CVD of 7.6% in men and women cancer survivors older than 30 yrs. More importantly, they also determined that the mean vascular age of cancer survivors was 8 years greater than their chronological age, suggesting that sub-clinical manifestation of CVD may be present within the vasculature of some cancer survivors.

The definition and scientific study of cardiotoxicity has, to date, primarily focused solely on the myocardial injury related to adjuvant cancer therapy and the National Cancer Institute has defined it as "toxicity that affects the heart" (http://www.cancer.gov/dictionary/). However, cancer survivors are also at risk for vascular-related abnormalities. Despite this risk, the impact of adjuvant treatments on the function and structure of the peripheral vascular system is still poorly understood. With normal aging, two of the most important vascular adaptations to arteries, which strongly contribute to the increased risk of vascular-related and general CVD, are an increase in large artery stiffness and dysfunction of the vascular endothelium [15, 16]. In subjects receiving anthracycline chemotherapy, Chaosuwannaki et al. (2010), Miza-Stec et al. (2013), and Draft et al. (2013) independently demonstrated significant increases in aortic stiffness 4-6 mo following treatment. Likewise, carotid intima-media thickness has been shown to increase within 6 mo of treatment with chemotherapy. This is critical given that arterial stiffness and intima-media thickness both are independently associated with increased risk of cardiovascular disease. In addition, carotid artery stiffness is a key determinant of the sympathetic baroreflex sensitivity in older men and women. This information suggests that decreases in baroreflex sensitivity may be occurring following chemotherapy treatment, which is important given it is a primary mechanism through which the autonomic nervous system regulates arterial blood pressure and that a low baroreflex sensitivity is associated with cardiovascular morbidity and mortality. Specific Aim 1 will address this question.

The vascular endothelium is the first physiological barrier encountered by intravenously administered chemotherapy. Unfortunately, the effects of adjuvant therapy on endothelial function have primarily been studied in childhood cancer survivors or following a single treatment session. Chow et al. (2006) observed a decreased brachial artery flow-mediated dilation (FMD), a measurement of endothelial-dependent dilation, ≈20 mo following anthracycline-based chemotherapy. Similarly, Vaughn et at. (2008) demonstrated a decreased FMD in long-term survivors of testicular cancer. In addition, several reports have demonstrated a decrease in arterial reactivity to various biological vasodilators (e.g., sodium nitroprusside, acetylcholine) following acute chemotherapy and radiation. In contrast to these studies, Jones et al. (2007) reported no difference in FMD in breast cancer patients ≈20 mo post-treatment compared to healthy controls. Increasing our understanding of the effects of chemotherapy on endothelial function is essential, especially since it can be the initial step in the development of cardiovascular disease.

Recently, the skin microcirculation has been used as a model circulation to evaluate the changes in vascular health in a variety of diseases including hypertension, renal disease, diabetes, atherosclerosis, coronary artery disease, and heart failure. This work has been facilitated, in part, by its easy accessibility and high responsiveness to biological vasodilators. Given the paucity of information on endothelial health in cancer patients undergoing anthracycline chemotherapy evaluation of the skin microcirculation provides a non-invasive and useful method of increasing our understanding of cardiotoxicity. Specific Aim 2 will address this problem.

Specific Aim 1: Evaluate the changes in spontaneous blood pressure control and arterial stiffness in patients treated with anthracycline-based chemotherapy.

Hypothesis 1a: Spontaneous baroreflex sensitivity will be significantly decreased in cancer patients and cancer survivors treated with anthracycline-based chemotherapy.

Hypothesis 1b: Changes in baroreflex control of blood pressure will be related to increases in carotid artery stiffness and cardiac changes in left ventricular ejection time.

Specific Aim 2: Evaluate the changes in macrovascular and microvascular vascular function.

Hypothesis 2a: Treatment with anthracycline-based chemotherapy will significantly decrease endothelium-dependent vasodilation in both the large brachial artery and the small microvascular capillaries in the skin.

Hypothesis 2b: Changes in vascular function will be associated with molecular markers of endothelial function and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study
* (Group 1) Diagnosed Stage I-III breast cancer or lymphoma cancer with a > 2 year life expectancy
* (Group 1) Current chemotherapy treatment includes anthracyclines
* (Group 2) History of Stage I-III breast cancer or lymphoma cancer with a > 2 year life expectancy
* (Group 2) 1 - 5 years removed from last date of anthracycline-based chemotherapy

Exclusion Criteria:

* History of clinical cardiovascular disease (Atherosclerotic cardiovascular disease (ASCVD) defined by history of acute coronary syndromes, myocardial infarction (MI), stable or unstable angina, coronary or other arterial revascularization, stroke, transient ischemia attack (TIA), or peripheral arterial disease presumed to be of atherosclerotic origin)
* Not met the above criteria
* Unable to provide informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer and lymphoma patients (n =20) will enter the study following completion of at least 1 cycle of chemotherapy. Breast cancer and lymphoma survivors (n=20) will enter study if they are 1 - 5 years removed from last date of chemotherapy. Healthy control subjects (n=20) will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Spontaneous baroreflex sensitivity | 1 day
  Measured once in each experimental group
Acetylcholine induced cutaneous (skin) blood flow (%) | 1 day
  Measured once in each experimental group

SECONDARY OUTCOMES:
Carotid artery stiffness | 1 day
  Measured once in each experimental group
Brachial-artery flow-mediated dilation | 1 day
  Measured once in each experimental group

CONTACTS AND LOCATIONS:
Locations (1):
- Lafene Health Center, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patnaik JL, Byers T, DiGuiseppi C, Dabelea D, Denberg TD. Cardiovascular disease competes with breast cancer as the leading cause of death for older females diagnosed with breast cancer: a retrospective cohort study. Breast Cancer Res. 2011 Jun 20;13(3):R64. doi: 10.1186/bcr2901. PMID 21689398
- [Background] Mulrooney DA, Blaes AH, Duprez D. Vascular injury in cancer survivors. J Cardiovasc Transl Res. 2012 Jun;5(3):287-95. doi: 10.1007/s12265-012-9358-7. Epub 2012 Mar 29. PMID 22456863
- [Background] Chaosuwannakit N, D'Agostino R Jr, Hamilton CA, Lane KS, Ntim WO, Lawrence J, Melin SA, Ellis LR, Torti FM, Little WC, Hundley WG. Aortic stiffness increases upon receipt of anthracycline chemotherapy. J Clin Oncol. 2010 Jan 1;28(1):166-72. doi: 10.1200/JCO.2009.23.8527. Epub 2009 Nov 9. PMID 19901105
- [Background] Duquaine D, Hirsch GA, Chakrabarti A, Han Z, Kehrer C, Brook R, Joseph J, Schott A, Kalyanaraman B, Vasquez-Vivar J, Rajagopalan S. Rapid-onset endothelial dysfunction with adriamycin: evidence for a dysfunctional nitric oxide synthase. Vasc Med. 2003 May;8(2):101-7. doi: 10.1191/1358863x03vm476oa. PMID 14518612
- [Background] Didier KD, Ederer AK, Reiter LK, Brown M, Hardy R, Caldwell J, Black C, Bemben MG, Ade CJ. Altered Blood Flow Response to Small Muscle Mass Exercise in Cancer Survivors Treated With Adjuvant Therapy. J Am Heart Assoc. 2017 Feb 7;6(2):e004784. doi: 10.1161/JAHA.116.004784. PMID 28174169
- [Background] Ederer AK, Didier KD, Reiter LK, Brown M, Hardy R, Caldwell J, Black CD, Larson RD, Ade CJ. Influence of Adjuvant Therapy in Cancer Survivors on Endothelial Function and Skeletal Muscle Deoxygenation. PLoS One. 2016 Jan 25;11(1):e0147691. doi: 10.1371/journal.pone.0147691. eCollection 2016. PMID 26807572